CLINICAL TRIAL: NCT04316247
Title: Demographic, Clinicopathological Characteristics and Survival of Breast Cancer Patients in Assiut University Hospital (2015-2019).
Brief Title: Demographic , Clinicopathological Characteristics and Survival of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Neveen Nageh Kamel Shalaby, Principal investigator, Assiut University
Other Study IDs: Neveen
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will retrospectively study the demographic , clinicopathological characteristics and survival of breast cancer patients admitted to Assiut University hospital from the year 2015 to 2019

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies in females, which is the second leading cause of cancer death throughout the world after lung cancer . The incidence of breast cancer has been increasing over the past decades , especially in young women (≤ 35 years old). There is approximately 182,000 women with breast neoplasm annually in the United States, accounting for about 26% of all incident cancers among women.

In Asia, the morbidity rate is as high as 9.5%-12% . Even worse in China, the average onset age of breast cancer might be 8-10 years younger than that in Western countries which account for upto 4% in total breast cancer patients .

In Egypt, breast cancer is the commonest type of female malignancy represented about 38.8% among common cancer sites in females.Although The unclear etiology of the majority of breast cancer, but there are numerous risk factors for the disease. Screening and early detection when combined with adequate, efficient treatment is considered the hope for a reduction of mortality in breast cancer as postulated by World Health organization (WHO).

ELIGIBILITY:
Inclusion Criteria:

* All histologically confirmed and documented patients with invasive ductal or lobular carcinoma of the breast attending at Assiut University hospital from year 2015 to 2019.

Exclusion Criteria:

* • Patients who previously received treatment outside Assiut University hospital.

  * A serious un controlled concomitant disease that would contraindicate with use of systemic treatment. .

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective study on breast cancer patients : A single institution study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The survival rate of breast cancer in assiut university hospital | One year
  The number of patients survived after surgery or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Samir E Shehata, Professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen S, Chen H, Yi Y, Jiang X, Lei H, Luo X, Chen Y, Liu S, Yuan D, Jia X, Li J. Comparative study of breast cancer with or without concomitant Paget disease: An analysis of the SEER database. Cancer Med. 2019 Jul;8(8):4043-4054. doi: 10.1002/cam4.2242. Epub 2019 May 28. PMID 31134761